CLINICAL TRIAL: NCT06506903
Title: Avalus Ultra Post-Approval Study (PAS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT23007
Record Dates: First submitted 2024-07-02; First posted 2024-07-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Avalus Ultra (Experimental): Avalus Ultra bioprosthesis: sizes 19mm, 21mm, 23mm, 25mm, 27mm, and 29mm
  Interventions: Device: Medtronic Avalus Ultra

INTERVENTIONS:
Device: Medtronic Avalus Ultra — Surgical aortic valve replacement with the Medtronic Avalus Ultra bioprosthesis for management of aortic stenosis and regurgitation.

SUMMARY:
The purpose of this study is to characterize the safety and effectiveness of the Medtronic Avalus Ultra aortic valve bioprosthesis in patients with aortic valve disease.

DETAILED DESCRIPTION:
A prospective, multi-center, single-arm, interventional, non-randomized, post-market study to characterize the safety and effectiveness of the Medtronic Avalus Ultra aortic valve bioprosthesis in patients with aortic valve disease. Approximately 150 subjects in the United States will be implanted and followed through one year post-procedure.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet the following criteria to be included in the study:

1. Subject has moderate or greater aortic stenosis or regurgitation, and there is a clinical indication for replacement of their native or prosthetic aortic valve with a bioprosthesis, with or without concomitant procedures, which are limited to any of the following:

   * Atrial fibrillation (AF) ablation
   * Ascending aortic aneurysm or dissection repair or replacement, with or without circulatory arrest
   * Coronary artery bypass graft (CABG)
   * Surgical management of the left atrial appendage (LAA)
   * Patent foramen ovale (PFO) closure
   * Resection of a sub-aortic membrane not requiring myectomy
2. Subject is geographically stable and willing to return to the implanting site for all follow-up visits
3. Subject is of legal age to provide informed consent
4. Subject has been adequately informed of risks and requirements of the study and is willing and able to provide informed consent for participation in the study

Exclusion Criteria

Subjects who meet any of the following criteria will not be eligible for participation in the study:

1. Subject has a pre-existing prosthetic valve or annuloplasty device in another position or requires replacement or repair of the mitral, pulmonary, or tricuspid valve
2. Subject has had a previous implant and then explant of the Avalus Ultra aortic valve bioprosthesis within the Avalus Ultra Post-Approval Study
3. Subject presents with active endocarditis, active myocarditis, or other systemic infection
4. Subject has a known hypersensitivity to contrast media that cannot be adequately premedicated
5. Subject has a known hypersensitivity to platinum, iridium, or tantalum
6. Subject has an anatomical abnormality that would increase surgical risk of morbidity or mortality, including:

   * Acute Type A aortic dissection
   * Ventricular aneurysm
   * Porcelain aorta
   * Hostile mediastinum
   * Hypertrophic obstructive cardiomyopathy
   * Documented pulmonary hypertension (systolic >60mmHg)
7. Subject has a non-cardiac major or progressive disease with a life expectancy of less than 1 year. These conditions include but are not limited to:

   * Child-Pugh Class C liver disease
   * Terminal cancer
   * End-stage lung disease
8. Subject has renal failure, defined by dialysis therapy or glomerular filtration rate (GFR) <30 mL/min/1.73 m2
9. Subject has active or untreated hyperparathyroidism
10. Subject is participating in another investigational device or drug trial (not including registries)
11. Subject is pregnant, lactating, or planning to become pregnant during the study period
12. Subject has a documented history of substance (drug or alcohol) abuse
13. Subject has greater than mild mitral valve regurgitation or greater than mild tricuspid valve regurgitation as assessed by echocardiography
14. Subject has systolic ejection fraction (EF) <20% as assessed by echocardiography
15. Subject has Grade IV diastolic dysfunction
16. Subject has documented bleeding diatheses
17. Subject has had an acute preoperative neurological deficit or myocardial infarction and has not returned to baseline or stabilized ≥30 days prior to implant
18. Subject requires emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Time-related incidence of adverse events and death through 1 year post-procedure | 30 days and 1 year post-procedure
  Safety of the valve is evaluated by the time-related incidence of valve-related adverse events and death. The following valve-related adverse events are evaluated in this study: thromboembolism, valve thrombosis, hemorrhage, paravalvular leak, endocarditis, structural valve deterioration, non-structural valve dysfunction, reintervention, death. This safety endpoint is descriptive, and no statistical hypothesis testing will be performed. The primary analysis of safety endpoint events will occur once all implanted participants have completed their 1 year post-procedure visit or exited the study.
Evaluation of Mean Pressure Gradient (mmHg) through 1 year post-procedure | 30 days and 1 year post-procedure
  Mean pressure gradient is evaluated by transthoracic echocardiography technique as the average flow of blood through the aortic valve measured in millimeters of mercury. This effectiveness endpoint is descriptive, and will be summarized as with continuous data. No statistical hypothesis testing will be performed. The primary analysis of effectiveness endpoint events will occur once all implanted participants have completed their 1 year post-procedure visit or exited.
Evaluation of Effective Orifice Area (cm^2) through 1 year post-procedure | 30 days and 1 year post-procedure
  Effective Orifice Area (EOA) is assessed by transthoracic echocardiography technique and is measured as the minimal cross-sectional area of the blood flow downstream of the aortic valve. This effectiveness endpoint is descriptive, and will be summarized as with continuous data. No statistical hypothesis testing will be performed. The primary analysis of effectiveness endpoint events will occur once all implanted participants have completed their 1 year post-procedure visit or exited.
Change in heart failure status based on NYHA functional classification from baseline through 1 year post-procedure | 30 days and 1 year post-procedure
  The change of the New York Heart Association (NYHA) functional classification at 30 days and 1 year from baseline will be used to evaluate the change heart failure status. The primary analysis will occur once all implanted participants have completed their 1 year visit or exited; no statistical hypothesis testing will be performed.
  Measure Description: Cardiac Disease with Functional Classes (lower value is more desirable than higher value) I - No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  II - Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  III - Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  IV - Symptoms of heart failure at rest. Any physical activity causes further discomfort.
Implanted valve size compared to pre-operative annulus dimensions on Multi-Detector Computed Tomography (MDCT) | 1 year post-procedure
  This effectiveness endpoint is descriptive, and no statistical hypothesis testing will be performed. The primary analysis of effectiveness endpoint events will occur once all implanted participants have completed their 1 year post-procedure visit or exited.
Characterization of post-operative stent deformation on Multi-Detector Computed Tomography (MDCT) | 1 year post-procedure
  This effectiveness endpoint is descriptive, and no statistical hypothesis testing will be performed. The primary analysis of effectiveness endpoint events will occur once all implanted participants have completed their 1 year post-procedure visit or exited.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Crestanello, MD, Principal Investigator — Mayo Clinic; Bo Yang, MD, PhD, Principal Investigator — University of Michigan
Locations (15):
- United States (15):
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida Shands, Gainesville, Florida
  - Emory Saint Joseph's, Atlanta, Georgia
  - WellStar Kennestone Hospital, Marietta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Michigan Health System - University Hospital, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Joseph's Hospital Health Center, Syracuse, New York
  - UH Cleveland Medical Center, Cleveland, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Heart Hospital of Austin, Austin, Texas
  - CHI Saint Lukes Health - Baylor Saint Lukes Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Swedish Medical Center Cherry Hill, Seattle, Washington